CLINICAL TRIAL: NCT07335263
Title: The Effect of Swaddling and Nesting Methods on Pain and Stress Levels in Newborns Undergoing Noninvasive Mechanical Ventilation
Brief Title: Effects of Swaddling and Nesting on Pain and Stress in Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025/01-29
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stress; Non Pharmacological Intervention; Newborn Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The focus of conducting a blinded clinical trial is to eliminate bias in participants, researchers, or those evaluating the results (Bhide et al., 2018). In this study, blinding of researchers is not possible because they personally performed the procedures in the study groups in the neonatal intensive care unit. The saliva samples collected in the study and other collected data will be blinded to both the ELISA technician and the statistician by assigning different group names.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swaddling Group (Experimental): Swaddling method, a soft-textured, 100% cotton, square-shaped (100×100 cm, 110 g) fabric blanket that does not irritate the newborn's skin will be used. The newborn will be placed on the blanket in a supine position, naked except for a diaper, with the top edge of the blanket aligned with the shoulders. The arms will be placed in an extension-adduction position and the upper body will be swaddled with the blanket. The lower section will be wrapped with the legs in flexion and abduction, leaving space at the bottom for the feet to move freely and ensuring that the wrapping is not too tight. The baby's head will be allowed to move freely.
  Interventions: Behavioral: Nesting
- Nesting Group (Experimental): Nesting method, swaddling devices covered with 100% cotton fabric, which support the intrauterine position and are routinely used in the neonatal intensive care unit, will be used. The swaddling device is confined with soft padding materials to support the baby's neck and body. The arms of the newborn placed in the supine position will be brought into the extension-adduction position and secured with soft elastic straps, and the baby's surroundings will be safely restricted. This method will ensure that the baby remains in a physiological and comfortable position.
  Interventions: Behavioral: swaddling

INTERVENTIONS:
Behavioral: swaddling — Saliva samples will be collected before the swaddling method is applied (t1), during application (5th minute) (t2), and 30 minutes after the swaddling method is applied (t3). Heart rate, respiratory rate, and partial oxygen pressure values, as well as pain and stress levels (ALPS-Neo), will be recorded by two researchers.
  Arms: Nesting Group
Behavioral: Nesting — Saliva samples will be collected before the nesting method is applied (t1), during application (5th minute) (t2), and 30 minutes after the nesting method is applied (t3). Heart rate, respiratory rate, and partial oxygen pressure values, as well as pain and stress levels (ALPS-Neo), will be recorded by two researchers.
  Arms: Swaddling Group

SUMMARY:
This study aims to investigate the effects of swaddling and cradling methods on pain and stress levels in newborn infants receiving respiratory support.

Infants receiving respiratory support in the neonatal intensive care unit may experience stress and discomfort during treatment. In this study, two different care methods that help infants feel more comfortable and secure will be scientifically compared. Only one of the Swaddling or Nesting methods will be applied to the newborns participating in the study. These methods are comfort-enhancing care practices routinely used in neonatal intensive care that do not harm the baby. The newborn's heart rate, respiratory rate, oxygen level, pain and stress symptoms will be closely and safely monitored by the healthcare team. A pain-free saliva sample will be collected to assess the newborn's stress level. It does not involve needles, does not hurt, and takes approximately 2 minutes. Pain and stress levels will be assessed in a multifaceted manner using clinical observation, physiological parameters, and saliva cortisol levels. The study aims to contribute to the strengthening of evidence-based non-pharmacological care practices in neonatal intensive care.

DETAILED DESCRIPTION:
This study was designed to investigate the effect of swaddling and nesting methods on pain and stress levels in newborns receiving nasal CPAP. The study was planned to be randomized and experimental in nature. The study population will consist of all newborns requiring nasal CPAP/noninvasive mechanical ventilation in the neonatal intensive care unit of a city hospital. The study will consist of two intervention groups. A total of 100 newborn patients (Swaddling group = 50, Nesting group = 50) will be included in the study after obtaining consent from the parents of newborns diagnosed with transient tachypnea, born at 35 weeks of gestation or older, who are receiving nasal CPAP/noninvasive mechanical ventilator treatment in the NICU and meet the inclusion criteria of the study. Environmental conditions that could cause stress to newborns (noise, heat, lighting, etc.) will be kept at optimal levels. When placed on nCPAP, the infant will be placed in the supine position to better observe chest movements and breathing patterns. To ensure the patency of the infant's airway, a slight extension position will be achieved using neck rolls. Respiratory distress in newborns receiving nCPAP, stress due to positive air pressure, and pain caused by the pressure of the nasal cannula on the nostrils will be assessed by two researchers using the ALPS-Neo Neonatal Pain and Stress Assessment Scale (ALPS-Neo). In the swaddling group, saliva samples will be collected before the swaddling method is applied (t1), during application (t2), and 30 minutes after the swaddling method is applied (t3). Heart rate, respiratory rate, partial oxygen pressure values, pain and stress levels (ALPS-Neo) will be recorded by two researchers. In the Nesting Group, saliva samples will also be collected before the Nesting method is applied (t1), during application (t2), and 30 minutes after the wrapping method is applied (t3). Heart rate, respiratory rate, partial oxygen pressure values, pain and stress levels (ALPS-Neo) will be recorded by two researchers. The saliva sample collection process will be performed by removing the cotton roll from the inner tube and holding it by one end under the baby's tongue or in the corners of the mouth (2.5 cm) where saliva can be collected for approximately 2 minutes until the cotton is thoroughly saturated with saliva (0.012-3.000 ug/dL). The roll of cotton will be held by its dry end and the wet part will be placed back into the inner tube, the tube cap will be closed, and barcodes with the patient's name written on them will be affixed to each sample taken. The collected saliva samples will be numbered and stored at -20°C in the refrigerator in the neonatal intensive care unit. On the same day, they will be transferred to the research laboratory (KUYAM) under cold chain conditions with research permission, and the sample size in the study groups will be completed. They will be stored at -80°C until the ELISA study time. The saliva sample collection process will be performed by removing the cotton roll from the inner tube and holding it by one end under the baby's tongue or in the corners of the mouth (2.5 cm) where saliva can be collected for approximately 2 minutes until the cotton is thoroughly saturated with saliva (0.012-3.000 ug/dL). The entire ELISA study will be conducted at the Kütahya Health Sciences University Research Laboratory (KUYAM), and the collected samples will be blinded for the ELISA worker. Saliva samples will be centrifuged again at 1000 g for 2 minutes to remove mucins and other particulate matter that could interfere with antibody binding and affect the results. When all samples have reached room temperature, pipette 25 μL of standard and sample into each well of the 96-well plate included in the kit. Next, add 200 μL of assay diluent to the 96-well plate using a micropipette and incubate at room temperature for 1 hour at 500 rpm. After incubation is complete, wash 4 times with 300 μL of wash buffer. After washing is complete, add 200 μL of TMB Substrate Solution to each well containing the sample and standards and incubate at room temperature in the dark at 500 rpm for 25 minutes. After the incubation process is complete, 50 μL of reaction stop solution will be added to each well. At this point, the reaction in the wells will be observed to turn from green to yellow, and after all wells have turned yellow, a spectrophotometric measurement will be made at a wavelength of 450 nm. Total concentrations will be calculated from the absorbance values for standards and samples, and cortisol levels will be reported in μg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Birth week greater than 35 weeks and birth weight greater than 2000 grams
* Requirement for nasal CPAP/noninvasive mechanical ventilation
* Legal guardians' consent to participate in the study
* Postnatal diagnosis of transient tachypnea of the newborn

Exclusion Criteria:

Mother:

* Taking cortisol-containing medication during the antenatal period
* Taking narcotics during the antenatal period
* Having chorioamnionitis
* Having a metabolic disorder (adrenal insufficiency, etc.)

Newborn:

* Amniotic fluid stained with meconium
* Being intubated
* Having an Apgar score below 6
* Receiving analgesic or narcotic drugs for sedation
* The newborn receiving cortisol-containing medication
* Being unable to obtain a saliva sample or the sample being contaminated with blood
* Signs of nasal injury during noninvasive mechanical ventilation
* Congenital defects (spina bifida, gastroschisis, etc.) that prevent positioning using the swaddling or cradling methods
* Resuscitation
* Cerebral hypoxia-ischemia
* Non-respiratory causes (congenital pneumonia, respiratory distress syndrome, congenital heart disease, hypocalcemia, persistent hypoglycemia, development of sepsis)
* Hypocalcemia (low calcium level detected in blood gas sample taken while establishing an intravenous line prior to nCPAP)

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Determining pain and stress scores in newborns based on measurement times | before swaddling and nesting (t1), during application (5th minute) (t2), and 30 minutes after the swaddling and nesting method was applied (t3)
  The ALPS-Neo Neonatal Pain and Stress Assessment Scale (ALPS-Neo) score was recorded by the researcher before swaddling and nesting (t1), during application (5th minute) (t2), and 30 minutes after the swaddling and nesting method was applied (t3). The ALPS-Neo is a 3-point Likert-type scale consisting of 5 items: the newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made through observation. As the score increases, stress and pain increase. The assessment results indicate that a score of 3-5 points indicates mild pain and stress, while a score above 5 points indicates severe pain and stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No